CLINICAL TRIAL: NCT06803030
Title: A Comparative Study on the Efficacy of Tamsulosin, Solifenacin and Mirabegron in Alleviating Ureteral Stent-related Symptoms: a Randomized Controlled Trial
Brief Title: Study of Tamsulosin, Solifenacin and Mirabegron in Alleviating Ureteral Stent-related Symptoms
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bir Hospital (Other Government)
Collaborators: Nepal Health Research Council (Other Government)
Responsible Party: Principal Investigator, Jainendra Kumar Manoj, M Ch Urology Resident, Bir Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BirH
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Ureteral Stent-Related Symptom
Keywords: Mirabegron; Tamsulosin; Solifenacin
MeSH Terms: interventions — Tamsulosin; Solifenacin Succinate; mirabegron

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Tamsulosin group (Active Comparator): placement of ureteral stents followed by Cap. Tamsulosin 0.4 mg once daily, to relieve the symptom
  Interventions: Drug: Tamsulosin Hydrochloride 0.4 mg
- Solifenacin group (Active Comparator): placement of ureteral stents followed by Tab Solifenacin 5 mg once daily, to relieve the symptom
  Interventions: Drug: Solifenacin Succinate 5 mg
- Mirabegron group (Active Comparator): placement of ureteral stents followed by Tab. Mirabegron 25 mg once daily, to relieve the symptom
  Interventions: Drug: Mirabegron 25 mg

INTERVENTIONS:
Drug: Tamsulosin Hydrochloride 0.4 mg — placement of ureteral stents followed by Cap. Tamsulosin 0.4 mg once daily
  Other Names: Cap. Urimax 0.4 mg
  Arms: Tamsulosin group
Drug: Solifenacin Succinate 5 mg — placement of ureteral stents followed by Tab. Solifenacin 5 mg once daily
  Other Names: Tab. Solay 5 mg
  Arms: Solifenacin group
Drug: Mirabegron 25 mg — placement of ureteral stents followed by Tab. Mirabegron 25 mg once daily
  Other Names: Tab. Mirasin 25 mg
  Arms: Mirabegron group

SUMMARY:
A comparative study on the efficacy of Tamsulosin, Solifenacin and Mirabegron in alleviating ureteral stent-related symptoms: a randomized controlled trial.

DETAILED DESCRIPTION:
Ureteral stent related symptoms can be a major issue in patient undergoing stent placement after any procedure such as- complains of pain, urinary symptoms, sex related and work related and other symptoms. These symptoms can be alleviated with use of drugs such as Tamsulosin, Solifenacin and Mirabegron. Patient recruited in each arm of the study will have their stent related symptoms scoring done using a validated outcome assessment tool to measure the ureteral stent-related symptoms, Ureteral Stent Symptom Questionnaire (USSQ) on day 1, day 7 and day 14 after the stent placement.

ELIGIBILITY:
Inclusion Criteria:

• Eligible participants were adult patients (aged 19-80 years) who underwent unilateral retrograde rigid ureteroscopy (URS) or retrograde intrarenal surgery (RIRS) with planned ureteric stent insertion for urinary tract stones

Exclusion Criteria:

* Concomitant use of a-blockers, anticholinergics, corticosteroids, calcium channel blockers, and analgesics
* Undergoing percutaneous nephrolithotomy, open ureteric surgery or laparoscopic ureteric surgery, including ureterolithotomy
* Neurogenic bladder, Over Active Bladder (OAB) syndrome, and neurological and psychiatric diseases
* Preoperative febrile Urinary Tract Infection (UTI)
* Pregnancy or breastfeeding;
* A single kidney
* Moderate or severe cardiovascular or cerebrovascular disease
* Hepatic dysfunction
* History of pelvic surgery or irradiation
* History of bladder or prostate surgery
* Other acute medical conditions (including acute pancreatitis, acute gastroenteritis, musculoskeletal disorders) that might influence the Ureteral Stent Symptom Questionnaire(USSQ) pain score
* Allergy to any medication

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Estimated)
Dates: Start 2025-08-30 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
alleviating Ureteral stent related symptoms | 2 weeks
  mitigating the ureteric stent related symptoms using structured questionnaire

SECONDARY OUTCOMES:
early removal of ureteral stent | before 2 weeks
  early removal of stent due to stent migration, fever, urosepsis

CONTACTS AND LOCATIONS:
Locations (1):
- NAMS, Bir Hospital, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No